CLINICAL TRIAL: NCT00002117
Title: A Randomized, Open-Label Study of Alternative Treatment Combinations of Dideoxycytidine (HIVID; ddC) and Zidovudine (AZT) in Patients With HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 220A; NV 14257
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-02

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To investigate the appropriate zalcitabine ( dideoxycytidine; ddC ) dose and zidovudine ( AZT ) schedule for use in combination therapy in patients with HIV infection.

DETAILED DESCRIPTION:
Patients are randomized to one of four treatment arms. ddC is administered at 1 of 2 doses every 8 hours. AZT is administered at 1 of 2 doses (every 4 hours while awake or every 8 hours).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 count 100 - 500 cells/mm3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Kaiser Foundation Hosp, Harbor City, California
  - Kaiser Permanente Med Ctr, Los Angeles, California
  - Sharp Rees - Stealy Med Group, San Diego, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Denver Public Health Dept / Disease Control Services, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Intergrated Care Ctr, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - New England Med Ctr, Boston, Massachusetts
  - St Paul Ramsey Med Ctr / HIV Program Office, Saint Paul, Minnesota
  - Washington Univ, St Louis, Missouri
  - Univ of New Mexico School of Medicine, Albuquerque, New Mexico
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Bronx Veterans Affairs Med Ctr, The Bronx, New York
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Oregon Health Sciences Univ, Portland, Oregon
  - N Texas Ctr for AIDS & Clin Rsch, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Dr Brian Buggy, Milwaukee, Wisconsin